CLINICAL TRIAL: NCT01241812
Title: Biomarkers and Knee Osteoarthritis: Associations With Joint Load and Effects of Exercise
Brief Title: Biomarkers and Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Arthritis Network (Network)
Responsible Party: Principal Investigator, Michael Hunt, Director, Motion Analysis and Biofeedback Lab, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H10-01492
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Knee Osteoarthritis
Keywords: knee; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A. (Experimental): 10 weeks of partially supervised lower limb muscle strengthening targeting the following muscles groups: quadriceps, hamstrings, hip abductors.
  Interventions: Behavioral: Lower limb muscle strengthening
- B (No Intervention)

INTERVENTIONS:
Behavioral: Lower limb muscle strengthening — Participants in the exercise group will receive a lower limb strengthening program consisting of 6 exercises targeting the quadriceps, hamstrings, and hip abductor groups. They will perform these exercises at home 4 times per week (3 sets of 10 repetitions per exercise). Over the course of the intervention, each participant will consult with the physiotherapist a total of 5 times (once per week in weeks: 1,2,3,5, and 8) to ensure proper performance of exercises and safe progression of resistance.
  Arms: A.

SUMMARY:
High joint load during walking has been linked to cartilage degradation. Biomarkers, found in the blood and urine, are protein fragments released after cartilage degradation characteristic of OA. They have the potential to enable direct and immediate disease state monitoring and identification of early cartilage changes. Little is known about the association of biomarkers with joint load or if exercise aimed at reducing joint load changes biomarker levels, thus reducing the risk of OA progression. This study will provide novel information on these relationships and will guide future intervention studies. The investigators hypothesize that certain biomarkers will be highly correlated with joint loading during walking and that the levels of these biomarkers in the blood and urine will decrease following an exercise intervention aimed at cartilage unloading.

DETAILED DESCRIPTION:
Participants will be tested twice (baseline and 11 weeks later) where they will undergo gait and strength analyses by the same blinded assessor, complete self-report questionnaires, and have blood and urine samples drawn. Participants will then be randomized into either: (i) exercise; or (ii) usual care (no additional treatment). Those in the exercise group will complete 10-weeks of strengthening targeting lower limb muscles. Once weekly, they will consult with the study physiotherapist (MAH) at UBC to ensure proper performance and safe progression of exercises. Participants will be given cuff weights and resistance bands to complete exercises at home five times per week. Exercise compliance will be monitored using log books. All participants will be encouraged to maintain their usual treatment regimen (except for exercises completed by the exercise group), but will document any unexpected alterations such as medication changes or physician visits.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 50 years (to meet the American College of Rheumatology clinical definition of OA)
* radiographically confirmed knee OA in the medial compartment of the tibiofemoral joint
* knee pain during walking greater than 3/10 (based on an 11-point scale; 0 = "no pain", 10 = "maximal pain") on most days of the previous month
* predominance of pain/tenderness over the medial (inside) region of the knee

Exclusion Criteria:

* articular cartilage degradation in the lateral tibiofemoral compartment greater than the medial (medial compartment OA is more common than lateral and the KAM is a validated measure of medial compartment loading only)
* currently in a structured exercise program
* medical condition precluding exercise
* inflammatory arthritic condition
* history of knee replacement surgery
* recent use of corticosteroids (oral or via injection)
* unable to attend exercise training sessions at UBC
* pain originating predominantly from the patellofemoral joint
* inability to ambulate without a gait aid
* non-English speaking (questionnaires are in English and must be completed by the study participant only)
* recent (within 6 months) arthroscopic knee surgery
* significant hip or back pain (limits the ability to perform the testing and exercises)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Serum levels of biomarkers (COMP, HA, C2C, CP2) measured at baseline and 11 weeks | 11 weeks
Urinary levels of biomarkers (CTX-2, C2C) measured at baseline and 11 weeks | 11 weeks

SECONDARY OUTCOMES:
Knee joint loading during walking (external knee adduction moment) measured at baseline and 11 weeks | 11 weeks
Self-reported pain and physical function (WOMAC) measured at baseline and 11 weeks. | 11 weeks
Isometric muscle strength (hamstrings, quadriceps, hip abductors) measured at baseline and 11 weeks | 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Hunt, PT, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Hunt MA, Pollock CL, Kraus VB, Saxne T, Peters S, Huebner JL, Sayre EC, Cibere J. Relationships amongst osteoarthritis biomarkers, dynamic knee joint load, and exercise: results from a randomized controlled pilot study. BMC Musculoskelet Disord. 2013 Mar 27;14:115. doi: 10.1186/1471-2474-14-115. PMID 23530976